CLINICAL TRIAL: NCT03632395
Title: Early Detection of Postoperative Anastomotic Leak by CT
Status: Completed | Type: Observational
Sponsor: BIRENDRA KUMAR SAH (Other)
Responsible Party: Sponsor-Investigator, BIRENDRA KUMAR SAH, Surgeon, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Other Study IDs: RJ-GC Postop-complication 1
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2018-08

CONDITIONS: Anastomotic Leak
Keywords: gastric cancer; postoperative complication; anastomotic leak; oral contrast agent; computed tomography
MeSH Terms: conditions — Anastomotic Leak; Stomach Neoplasms; Postoperative Complications | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: computed tomography — computed tomography

SUMMARY:
Postoperative anastomotic leak is rare but life threatening complication after gastric cancer surgery. Early diagnosis is key to minimize other hazards which are caused by anastomotic leak. Investigators introduced a novel method to detect early diagnosis of anastomotic leak after gastric cancer surgery.

DETAILED DESCRIPTION:
Postoperative anastomotic leak is rare but life threatening complication after gastric cancer surgery. Early diagnosis is key to minimize other hazards which are caused by anastomotic leak. Investigators introduced a novel method to detect early diagnosis of anastomotic leak after gastric cancer surgery. Oral contrast agent is used for CT. Investigators carefully collected all the data prospectively and standard definition of anastomotic leak was applied.

ELIGIBILITY:
Inclusion Criteria:

Patients with gastric cancer surgery

Exclusion Criteria:

Patients with non gastric cancer surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent gastric cancer surgery.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of anastomotic leak | 5-10 days after surgery
  CT was routinely used to detect early anastomotic leak after gastric cancer surgery

CONTACTS AND LOCATIONS:
Overall Officials: BIRENDRA K SAH, Ph D, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China